CLINICAL TRIAL: NCT05907226
Title: Conducting a Study to Compare Smokers' Appraisal of Proposed Plain Packs and Existing Cigarette Packs in Hong Kong
Brief Title: Compare Smokers' Appraisal of Proposed Plain Packs and Existing Cigarette Packs
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Other Study IDs: NTEC-2023-179
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Health Risk Behaviors; Non Communicable Diseases
Keywords: Plain cigarette packs; current smokers; branded cigarette packs
MeSH Terms: conditions — Health Risk Behaviors; Noncommunicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
2 Objectives

1. To explore the noticeability of pictorial health warnings and perceptions of attractiveness and harmfulness towards plain cigarette packets and existing cigarette packets with 85% pictorial warnings in current smokers;
2. to compare the differences in perceptions of packaging in current smokers with different characteristics (i.e. by sex, age, the consumption level of cigarettes, nicotine dependence levels, and types of tobacco used for polytobacco product users);
3. to evaluate the effectiveness in reducing smoking consumption and promoting quit attempts; and
4. to assess the support for the legislation of plain packaging.

DETAILED DESCRIPTION:
The present study will recruit at least 1,280 current smokers at smoking hotspots in Hong Kong Island, Kowloon, and the New Territories. Land-based, non-institutionalized Hong Kong residents aged 18 years and over who speak Cantonese or Putonghua are eligible to participate.

Subjects will be shown dummies of branded and plain packets that differ in brand names and plain colours. Subjects will discuss their perceptions of attractiveness and harmfulness, noticeability of warnings and effectiveness in reducing smoking consumption and promoting quit attempts. Their opinions on the legislation of plain packaging will also be asked.

After each interview, interviewers will debrief each interviewee on the harms of smoking and distribute a card providing a quitline and quitting methods.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 years and over
* Able to speak Cantonese or Putonghua
* Smokers who have tobacco use behaviour of holding a cigarette in the hand or mouth

Exclusion Criteria:

* Foreign domestic helpers
* Non-smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 1,280 current smokers at smoking hotspots in Hong Kong Island, Kowloon, and the New Territories will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 1283 (Actual)
Dates: Start 2023-06-04 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Percent of participants who perceive current branded packets as attractive | Baseline
  Perceived attractiveness towards existing cigarette packets with 15 percent brand logo
Percent of participants who perceive plain packets as harmful | Baseline
  Perceived harmfulness towards plain packets

SECONDARY OUTCOMES:
Noticeability of pictorial warnings | Baseline
  Noticeability of pictorial warnings of plain cigarette packets and existing cigarette packets with 85% pictorial warnings in current smokers will be compared
Perceived effectiveness | Baseline
  The effectiveness in reducing smoking consumption and promoting quit attempts

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — williamli@cuhk.edu.hk
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No